CLINICAL TRIAL: NCT06854848
Title: Cohort of Patients With Systemic Granulomatosis (Sarcoidosis and Other Systemic Granulomatoses) and Associated Biological Collection GRAMI-BIO Study
Brief Title: Cohort of Patients With Systemic Granulomatosis and Associated Biological Collection
Acronym: GRAMI-BIO
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2024/73
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Granulomatosis
Keywords: Granulomatosis; sarcoidosis; Biological collection
MeSH Terms: conditions — Sarcoidosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 30 ml whole blood for Peripheral blood mononuclear cell (PBMC) and monocytes isolation and 10 ml urine sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Granulomatosis
  Interventions: Biological: blood sample; Biological: urine sample

INTERVENTIONS:
Biological: blood sample — 30 ml whole blood for Peripheral blood mononuclear cell (PBMC) and monocytes isolation
Biological: urine sample — 10 ml

SUMMARY:
The GRAMI-BIO study is a prospective single-centre cohort study to recruit 150 patients followed up in the the Bordeaux University Hospital. The total duration of the GRAMI-BIO study is ten years (five years of inclusion with five years of follow-up): Consecutive inclusion of patients meeting the definition of systemic granulomatosis. The main objective of this cohort is to describe to clinical progression of systemic granulomatosis and to collect blood fraction samples (serum bank, plasma bank, urine bank, DNA bank) from subjects participating in the cohort.

DETAILED DESCRIPTION:
Systemic granulomatosis is a group of diseases whose common feature is the anatomopathological existence of giganto-cellular granulomas composed of macrophages, epithelial cells and CD4+ T lymphocytes. The exact cause of the development of these granulomas remains unknown, although numerous studies suggest the hypothesis of environmental factors (infectious, exposure to particles) and genetic susceptibility factors. The persistence of granulomas is deleterious, ultimately leading to local destruction and tissue damage resulting in fibrosis of neighbouring tissues. Granulomatosis is a heterogeneous group in terms of aetiology: schematically, either an aetiology is identified: infection, environmental factors (berylliosis, pneumoconiosis), iatrogenesis (drugs), neoplasia, immune deficiency; or granulomatosis is said to be idiopathic, the most common case, falling within the definition of systemic sarcoidosis. Therefore, with a view to future research work, it seems imperative to set up a biological bank of patients being monitored for systemic granulomatosis within the division. It is particularly important to identify genetic variants, circulating biomarkers associated with the onset, severity and response to treatment of these diseases. The main aim of the "GRAMI-BIO" study is to describe the clinical evolution of patients with systemic granulomatosis (sarcoidosis and other granulomatoses) followed at the Bordeaux University Hospital, and to collect samples from blood fractionation (serum bank, plasma bank, urine bank, DNA, RNA bank) to constitute a biobank.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or over
* Patients with systemic granulomatosis (diagnosis proven by anatomopathological sampling) at diagnosis.
* Persons affiliated to or benefiting from a social security scheme.
* Free, informed and written consent signed by the participant and the investigator (at the latest on the day of inclusion and before any examination required by the research).

Exclusion Criteria:

* Patients infected with human immunodeficiency virus (HIV), Hepatitis B virus (HBV) and/or Hepatitis C virus (HCV)
* Pregnant or breast-feeding women
* Patients already receiving specific treatment for systemic granulomatosis
* Persons deprived of their liberty by a judicial or administrative decision, minors, persons of legal age who are the object of a legal protection measure or unable to express their consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with systemic granulomatosis (diagnosis proven by anatomopathological sampling)
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Describe the clinical progression of systemic granulomatosis | At baseline (Day 0) and 60 months after baseline

SECONDARY OUTCOMES:
Identify predictive factors for the progression of the disease | At baseline (Day 0) and 60 months after baseline
Identify the management methods into patients with systemic granulomatosis | At baseline (Day 0) and 60 months after baseline
Identify predictive factors for response to treatments | At baseline (Day 0) and 60 months after baseline
Identify new clusters of the disease in a large population both clinically and biologically | At baseline (Day 0) and 60 months after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel RIBEIRO, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux - service de Médecine Interne et Immunologie Clinique, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No